CLINICAL TRIAL: NCT04034966
Title: Utility of Telemedicine in the Follow-Up of Patients in Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R-2018-785-035
Record Dates: First submitted 2018-10-31; First posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Chronic Kidney Disease Stage 5; Peritoneal Dialysis Complication
Keywords: peritoneal dialysis; Claria; telemedicine
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The Project will consist in the conventional clinical treatment of the APD patient cared for in IMSS regarding the kind of dialysis solution, handling of laboratory and office procedures, as well as the handling of complications. One arm will utilize the Claria device, and the other will utilize normal treatment procedures.
  The APD device in the control group will be called Claria® (Baxter, S.A. de C.V.) without the telemedicine device, and in the intervention group it will be the same device with the telemedicine module. Handling will be done according to the basic operating instructions established by the manufacturer.
  According to the preliminary analysis of the flow of patients in PD indicated in the above paragraphs, recruitment of the sample size will not represent a problem. Infrastructure available in both technical and experienced human resources makes the study feasible.
Masking Description: 750 Patients will be cluster randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Claria (Active Comparator): The APD device in the control group will be called Claria® (Baxter, S.A. de C.V.) with the telemedicine module. The telemedicine module is the platform for storing patient information directly from the PD machine. Handling will be done according to the basic operating instructions established by the manufacturer.
  Interventions: Device: Claria telemedicine device
- Control (No Intervention): The APD device in the control group will be called Claria® (Baxter, S.A. de C.V.) without the telemedicine device. the device is used for automated peritoneal dialysis. Handling will be done according to the basic operating instructions established by the manufacturer.

INTERVENTIONS:
Device: Claria telemedicine device — Use of Claria telemedicine module, which stores patient information in the cloud.
  Arms: Claria

SUMMARY:
Peritoneal dialysis (PD) technology is available but has not been tested in the real world. Therefore, the aim of this study is to test the utility of telemedicine in reducing mortality, hospitalizations, unscheduled visits, and cost derived from preventable complications. Incident patients to PD treatment will be followed from various hospitals in Mexico City and Guadalajara. Direct medical costs will be evaluated, along with unplanned hospital visits and complications over 2 years using the Claria telemedicine apparatus from Baxter Laboratories.

DETAILED DESCRIPTION:
Study Background & Rationale: (background information including previous studies as applicable )

Chronic kidney disease (CKD) is a growing problem world-wide which increases in parallel with some risk factors such as chronic diseases, mainly diabetes mellitus and hypertension. CKD imposes elevated costs both from the standpoint of human resources and hospital infrastructure, and above all in the economic aspect. In the United States, the cost of CKD equals more than 30 billion USD a year to care for a population of 450,000 patients, which means an elevated cost per patient per year. Mexico does not have precise statistics but it is estimated that the burden of the disease is higher than that faced by other health institutions in any of the therapeutic modalities. For IMSS, chronic kidney disease is found among the six diseases that cause the greatest expenses, datum that is magnified when considering that the current population in any dialysis program consists of only 60,000 patients. On the other hand, the number of nephrologists is insufficient to care for the patients, considering that the proportion recommended is 100 patients per nephrologist in dialysis programs. In IMSS, these proportions are greatly surpassed, and the need to increase human resources or use alternative technologies to ease the task is evident.

Since its introduction at the end of the 70's, peritoneal dialysis (PD) has been consolidated in many countries as a viable, long-term substitutive therapy for renal function. Frequency of use of PD in patients with end-stage renal disease (ESRD) has broad variations, from zero in some regions of France and Japan to 40% in the United Kingdom, 60% in Mexico, and 80% in Hong Kong.

In terms of outcomes, PD and hemodialysis (HD) are comparable. Mortality in PD is similar and even less than in HD, and the greatest advantage of PD over HD is its home application and simplified technique, since it gives the patient total autonomy for daily life. This advantage is even greater with nocturnal automated systems, or automated PD (APD).

In recent years, the concept of "telemedicine" has been developed, term that is used to name all electronic transfers of data, audio and video between the health team and patients, with the purpose of consultation, examination or performing long-distance medical procedures.

The facility of electronic communication has empowered the advantages of PD; with the use of telemedicine systems the rate of hospitalization has been reduced from 5.7 to 2.2, resulting in lower costs. One worry behind these efforts is knowing if the patients are prepared to join these systems. Luckily, the results of some surveys indicate that the degree of acceptance is high.

Telemedicine systems applied to PD include telephone devices with connection to land phones, tablets or teleconferences via the network. In Japan, telemedicine is used to monitor blood pressure, heart frequency, urinary volume or serum glucose, and in Spain it has been used for teleconferences, for clinical visits and audiovisual presentations to re-train patients. In Canada, contact through tablets favored communication between patients and health staff and, through the introduction of alerts in structured interviews; a significant number of hospital visits were avoided. In addition, they obtained a high level of patient satisfaction with the system.

Even when APD is an effective, safe procedure for treating patients with ESRD, the nephrologist depends on an important number of data that the patient should offer in order to write a prescription adjusted to the clinical conditions of each case. Some very illustrative aspects are, for example:

1. Ultrafiltration and total liquid removal (dialysis + urine) are crucial data to prescribe osmolarity and glucose content in dialysate. According to the clinical practice guides, there should be a minimum volume of 1.0 L/day, without forgetting that each mL of ultrafiltration is associated with the absorption of an important amount of glucose, with the consequent metabolic cost.
2. The volume of infused liquid should be adjusted to the body surface area of the patient, and should take into account that the total volume in the peritoneum has an additional increase from the ultrafiltration obtained. This should be achieved without exceeding the patient's tolerance and without forcing the generation of inflammatory stimuli.
3. In general, treatment adherence is estimated by the monthly consumption of dialysis solutions and patient self-reporting. However, the two procedures contain a large amount of subjectivity.
4. Adjustment or prescription of automated peritoneal dialysis (APD) requires calculation of the effective time of presence of the solutions in the cavity; that is, from the start of infusion to the end of drainage, discounting transit time.

All these data are impossible to obtain in a nocturnal treatment without the support of telemedicine. One aspect of great importance comes from the lack of achieving prescription goals, which negatively impacts clinical outcomes and incurs additional costs for unscheduled doctor visits and treatment of complications that are preventable through closer follow-up, such as the case of fluid overload through lack of ultrafiltration and symptoms of uremic syndrome from insufficient dialysis.

Potentially preventable hospitalization is understood as hospitalizations caused by ambulatory handling. It is about clinical conditions that can be prevented with good handling externally and that are recognized as indicators of efficiency in ambulatory handling. For the case of this project, in which telemedicine is expected to help make dialysis and ultrafiltration more efficient, potentially preventable hospitalizations will be considered in manifestations of uremic syndrome, hyperkalemia, and those derived from liquid overload, such as: edema, hypertension and heart failure.

Before the impossibility of obtaining complete, objective information necessary for the prescription of APD and adequate management of the patient, APD machines have incorporated a telemedicine module that recovers information on movement and volume of dialysis solution, glucose concentration, and in addition to objectively measuring treatment adherence. This new technology is already available, but its use in the "real world" has not been evaluated. Having this information in the investigator's medium is necessary, given that PD treatment predominates, especially in IMSS, which is the institution on which the weight of ESRD in the country rests.

ELIGIBILITY:
Inclusion Criteria: Hospitals will be randomly assigned to control (without telemedicine device) or intervention groups (with telemedicine device). Hospitals will be selected and matched according their basic infrastructure (Outpatient dialysis clinic, Emergency Room, Laboratory and Radiology Departments, Hospitalization Facility, accessibility to the internet and direct telephone communication with the patient and/or contact or person in charge of the patient), as well as Human Resources (Nephrologist, Internist, specialists to attend to the most frequent complications of PD, Nurses trained in PD, and Social Workers), and availability of a structured PD Program (Manuals, Supervised training programs for patients and caregivers, Registers for peritonitis, technique failure, and mortality rates).

Inclusion criteria

* Over 18 years of age
* Diagnosed with chronic kidney disease
* Incident to automated peritoneal dialysis
* Agree to sign informed consent

Exclusion Criteria:

* seropositive for HIV, hepatitis B or C, with cancer
* in treatment with immunosuppressors or with acute complications in the 30 days previous to recruitment.
* patients who voluntarily withdraw from the study, who change residence or who lose social security coverage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
MORTALITY RATE | 2 years
  Number of patients who lose their lives for every 100 years / patient at risk. Deaths/100 years/patient at risk.
DAYS OF HOSPITALIZATION | 2 years
  Number of days in the hospital per 100 years / patient at risk. Days/100 years/patient at risk.
DAYS OF PREVENTABLE HOSPITALIZATION | 2 years
  Number of days in the hospital for causes that can be corrected with efficient PD for every 100 years / patient at risk. Days/100 years/patient at risk.

SECONDARY OUTCOMES:
COSTS | 2 years
  These are the costs of using necessary services with the provision of dialysis and associated complications and comorbidities.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Salamanca, PhD, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Unidad de Investigacion Medica en Enfermedades Nefrologicas, Hospital de Especialidades Centro Medico Nacional Siglo XXI, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levey AS, Atkins R, Coresh J, Cohen EP, Collins AJ, Eckardt KU, Nahas ME, Jaber BL, Jadoul M, Levin A, Powe NR, Rossert J, Wheeler DC, Lameire N, Eknoyan G. Chronic kidney disease as a global public health problem: approaches and initiatives - a position statement from Kidney Disease Improving Global Outcomes. Kidney Int. 2007 Aug;72(3):247-59. doi: 10.1038/sj.ki.5002343. Epub 2007 Jun 13. PMID 17568785
- [Background] Amato D, Alvarez-Aguilar C, Castaneda-Limones R, Rodriguez E, Avila-Diaz M, Arreola F, Gomez A, Ballesteros H, Becerril R, Paniagua R. Prevalence of chronic kidney disease in an urban Mexican population. Kidney Int Suppl. 2005 Aug;(97):S11-7. doi: 10.1111/j.1523-1755.2005.09702.x. PMID 16014087
- [Background] USRDS Annual Report 2015. Chapter 11: Medicare Expenditures for Persons with ESRD
- [Background] Cortes-Sanabria L, Paredes-Cesena CA, Herrera-Llamas RM, Cruz-Bueno Y, Soto-Molina H, Pazarin L, Cortes M, Martinez-Ramirez HR. Comparison of cost-utility between automated peritoneal dialysis and continuous ambulatory peritoneal dialysis. Arch Med Res. 2013 Nov;44(8):655-61. doi: 10.1016/j.arcmed.2013.10.017. Epub 2013 Nov 8. PMID 24211750
- [Background] Informe al Ejecutivo Federal y al Congreso de la Unión 2015-2016V.6.1. Análisis del gasto en enfermedades crónico-degenerativas de alto impacto financiero para el IMSS. El Consejo Técnico del Instituto Mexicano del Seguro Social. Ciudad de México, junio de 2016
- [Background] Harley KT, Streja E, Rhee CM, Molnar MZ, Kovesdy CP, Amin AN, Kalantar-Zadeh K. Nephrologist caseload and hemodialysis patient survival in an urban cohort. J Am Soc Nephrol. 2013 Oct;24(10):1678-87. doi: 10.1681/ASN.2013020123. Epub 2013 Aug 8. PMID 23929773
- [Background] Thomas-Hawkins C, Flynn L, Clarke SP. Relationships between registered nurse staffing, processes of nursing care, and nurse-reported patient outcomes in chronic hemodialysis units. Nephrol Nurs J. 2008 Mar-Apr;35(2):123-30, 145; quiz 131. PMID 18472681
- [Background] Balaskas EV, Ikonomopoulos D, Sioulis A, Dombros N, Kassimatis E, Bamichas G, Katsara I, Tourkantonis A. Survival and complications of 225 catheters used in continuous ambulatory peritoneal dialysis: one-center experience in Northern Greece. Perit Dial Int. 1999;19 Suppl 2:S167-71. PMID 10406512
- [Background] USRDS Annual Report 2015. Chapter 13: International Comparisons.
- [Background] Pecoits-Filho R, Campos C, Cerdas-Calderon M, Fortes P, Jarpa C, Just P, Luconi P, Lugon JR, Pacheco A, Paniagua R, Rodriguez K, Sanabria M, Sciaraffia V, Velasco C, De Arteaga J. Policies and health care financing issues for dialysis in Latin America: extracts from the roundtable discussion on the economics of dialysis and chronic kidney disease. Perit Dial Int. 2009 Feb;29 Suppl 2:S222-6. PMID 19270223
- [Background] Jiwakanon S, Chiu YW, Kalantar-Zadeh K, Mehrotra R. Peritoneal dialysis: an underutilized modality. Curr Opin Nephrol Hypertens. 2010 Nov;19(6):573-7. doi: 10.1097/MNH.0b013e32833d67a3. PMID 20639759
- [Background] Mehrotra R. Choice of dialysis modality. Kidney Int. 2011 Nov;80(9):909-911. doi: 10.1038/ki.2011.262. PMID 21997506
- [Background] Lukowsky LR, Mehrotra R, Kheifets L, Arah OA, Nissenson AR, Kalantar-Zadeh K. Comparing mortality of peritoneal and hemodialysis patients in the first 2 years of dialysis therapy: a marginal structural model analysis. Clin J Am Soc Nephrol. 2013 Apr;8(4):619-28. doi: 10.2215/CJN.04810512. Epub 2013 Jan 10. PMID 23307879
- [Background] Gallar P, Vigil A, Rodriguez I, Ortega O, Gutierrez M, Hurtado J, Oliet A, Ortiz M, Mon C, Herrero JC, Lentisco C. Two-year experience with telemedicine in the follow-up of patients in home peritoneal dialysis. J Telemed Telecare. 2007;13(6):288-92. doi: 10.1258/135763307781644906. PMID 17785025
- [Background] Nakamoto H, Nishida E, Ryuzaki M, Sone M, Yoshimoto M, Itagaki K. Blood pressure monitoring by cellular telephone in patients on continuous ambulatory peritoneal dialysis. Adv Perit Dial. 2004;20:105-10. PMID 15384807
- [Background] Edefonti A, Boccola S, Picca M, Paglialonga F, Ardissino G, Marra G, Ghio L, Parisotto MT. Treatment data during pediatric home peritoneal teledialysis. Pediatr Nephrol. 2003 Jun;18(6):560-4. doi: 10.1007/s00467-003-1147-8. Epub 2003 Apr 29. PMID 12720083
- [Background] Cargill A, Watson AR. Telecare support for patients undergoing chronic peritoneal dialysis. Perit Dial Int. 2003 Jan-Feb;23(1):91-4. No abstract available. PMID 12691517
- [Background] Ghio L, Boccola S, Andronio L, Adami D, Paglialonga F, Ardissino G, Edefonti A. A case study: telemedicine technology and peritoneal dialysis in children. Telemed J E Health. 2002 Winter;8(4):355-9. doi: 10.1089/15305620260507486. PMID 12626104
- [Background] Lew SQ, Sikka N. Are patients prepared to use telemedicine in home peritoneal dialysis programs? Perit Dial Int. 2013 Nov-Dec;33(6):714-5. doi: 10.3747/pdi.2012.00203. No abstract available. PMID 24335134
- [Background] Nakamoto H. Telemedicine system for patients on continuous ambulatory peritoneal dialysis. Perit Dial Int. 2007 Jun;27 Suppl 2:S21-6. PMID 17556306
- [Background] Gallar P, Gutierrez M, Ortega O, Rodriguez I, Oliet A, Herrero JC, Mon C, Ortiz M, Molina A, Vigil A. [Telemedicine and follow up of peritoneal dialysis patients]. Nefrologia. 2006;26(3):365-71. Spanish. PMID 16892826
- [Background] Dey V, Jones A, Spalding EM. Telehealth: Acceptability, clinical interventions and quality of life in peritoneal dialysis. SAGE Open Med. 2016 Oct 4;4:2050312116670188. doi: 10.1177/2050312116670188. eCollection 2016. PMID 27757228
- [Background] Avila-Diaz M, Ventura MD, Valle D, Vicente-Martinez M, Garcia-Gonzalez Z, Cisneros A, Furlong MD, Gomez AM, Prado-Uribe MD, Amato D, Paniagua R. Inflammation and extracellular volume expansion are related to sodium and water removal in patients on peritoneal dialysis. Perit Dial Int. 2006 Sep-Oct;26(5):574-80. PMID 16973513
- [Background] Paniagua R, Ventura MD, Avila-Diaz M, Hinojosa-Heredia H, Mendez-Duran A, Cueto-Manzano A, Cisneros A, Ramos A, Madonia-Juseino C, Belio-Caro F, Garcia-Contreras F, Trinidad-Ramos P, Vazquez R, Ilabaca B, Alcantara G, Amato D. NT-proBNP, fluid volume overload and dialysis modality are independent predictors of mortality in ESRD patients. Nephrol Dial Transplant. 2010 Feb;25(2):551-7. doi: 10.1093/ndt/gfp395. Epub 2009 Aug 12. PMID 19679559
- [Background] Paniagua R, Ventura Mde J, Rodriguez E, Sil J, Galindo T, Hurtado ME, Alcantara G, Chimalpopoca A, Gonzalez I, Sanjurjo A, Barron L, Amato D, Mujais S. Impact of fill volume on peritoneal clearances and cytokine appearance in peritoneal dialysis. Perit Dial Int. 2004 Mar-Apr;24(2):156-62. PMID 15119636
- [Background] Fischbach M, Issad B, Dubois V, Taamma R. The beneficial influence on the effectiveness of automated peritoneal dialysis of varying the dwell time (short/long) and fill volume (small/large): a randomized controlled trial. Perit Dial Int. 2011 Jul-Aug;31(4):450-8. doi: 10.3747/pdi.2010.00146. Epub 2011 Mar 31. PMID 21454393
- [Background] Ronksley PE, Hemmelgarn BR, Manns BJ, Wick J, James MT, Ravani P, Quinn RR, Scott-Douglas N, Lewanczuk R, Tonelli M. Potentially Preventable Hospitalization among Patients with CKD and High Inpatient Use. Clin J Am Soc Nephrol. 2016 Nov 7;11(11):2022-2031. doi: 10.2215/CJN.04690416. Epub 2016 Oct 6. PMID 27821636
- [Background] Paniagua R, Ramos A, Fabian R, Lagunas J, Amato D. Chronic kidney disease and dialysis in Mexico. Perit Dial Int. 2007 Jul-Aug;27(4):405-9. PMID 17602147